CLINICAL TRIAL: NCT05657431
Title: The Effect of Ylang Ylang Oil and Lemon Oil Inhalation on Active Phase Labor Pain and Anxiety in Primiparous Pregnant Women
Brief Title: The Effect of Ylang Ylang Oil and Lemon Oil
Acronym: Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem Çağan (Other)
Responsible Party: Sponsor-Investigator, Özlem Çağan, assistant professor, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Cagan01
Record Dates: First submitted 2022-11-11; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pain, Labor; Anxiety; Aromatherapy
Keywords: primiparous; labor pain; aromatherapy; lemon oil; ylang ylang oil
MeSH Terms: conditions — Labor Pain; Anxiety Disorders | interventions — Oils, Volatile; Sodium Chloride; lemon oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Ylang ylang oil) (Experimental): A square cotton ball impregnated with a drop of ylang-ylang oil was placed in the participants randomized to group I (cervical dilatation ≥ 5) with the help of safety pins of pregnant women. One hour after the intervention (in the range of 5-7 cm cervical dilatation), pain levels were measured again with the VAS and anxiety levels were measured with the State Anxiety Scale. The essential oil was renewed as 1 drop every hour until the birth of the baby. When cervical dilatation was in the range of 8-10 cm, pain level was re-evaluated only with VAS. Spielberger Continuity Anxiety Scale was applied with face-to-face interview technique within 4-24 hours following the birth.
  Interventions: Other: essential oils (Ylang ylang oil)
- group 2 (Lemon oil) (Experimental): A square cotton ball impregnated with a drop of lemon oil was placed in the participants randomized to group 2 (cervical dilatation ≥ 5) with the help of safety pins of pregnant women. One hour after the intervention (in the range of 5-7 cm cervical dilatation), pain levels were measured again with the VAS and anxiety levels were measured with the State Anxiety Scale. The essential oil was renewed as 1 drop every hour until the birth of the baby. When cervical dilatation was in the range of 8-10 cm, pain level was re-evaluated only with VAS. Spielberger Continuity Anxiety Scale was applied with face-to-face interview technique within 4-24 hours following the birth.
  Interventions: Other: essential oils (lemon oil)
- group 3 (Control) (Placebo Comparator): A square cotton ball impregnated with a drop of salin was placed in the participants randomized to group I (cervical dilatation ≥ 5) with the help of safety pins of pregnant women. One hour after the intervention (in the range of 5-7 cm cervical dilatation), pain levels were measured again with the VAS and anxiety levels were measured with the State Anxiety Scale. The essential oil was renewed as 1 drop every hour until the birth of the baby. When cervical dilatation was in the range of 8-10 cm, pain level was re-evaluated only with VAS. Spielberger Continuity Anxiety Scale was applied with face-to-face interview technique within 4-24 hours following the birth.
  Interventions: Other: placebo (saline solutions)

INTERVENTIONS:
Other: essential oils (Ylang ylang oil) — inhaler aromatherapy
  Arms: group 1 (Ylang ylang oil)
Other: placebo (saline solutions) — placebo saline solutions
  Arms: group 3 (Control)
Other: essential oils (lemon oil) — inhaler aromatherapy
  Arms: group 2 (Lemon oil)

SUMMARY:
This study was conducted as a randomized controlled experimental study.To evaluate the effects of aromatherapy, one of the non-pharmacological pain methods, on labor pain and anxiety in the active phase in primiparous pregnant women.

The main questions it aims to answer are:

Is ylang ylang oil applied as an inhaler effective in reducing labor pain and anxiety? Is lemon oil applied as an inhaler effective in reducing labor pain and anxiety? Participants randomized according to the closed envelope method into the lemon oil group (n=15), ylang ylang oil group (n=15) and control group (n=15). In the active phase (cervical dilatation ≥5), a drop of essential oil was instilled onto square cotton balls to the intervention groups and renewed as one drop every hour until labor occurred. In the control group, 1 drop of saline was dripped onto square cotton balls. Visual pain scale (VAS) and state anxiety ınventory were applied to the intervention groups and control groups before the application. After the application, VAS and state anxiety ınventory were evaluated at 5-7 cm dilatation, and only with VAS at 8-10 cm dilatation. The trait anxiety ınventory was administered to the volunteers after birth.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (37-41 weeks)
* Pregnant women between the ages of 18-35
* had singleton pregnancy with cephalic presentation of the fetus
* Not allergic to ylang ylang oil, flower/lemon or oil or anything
* Absence of any pregnancy complications
* No previous miscarriage, no abortion
* Not having any diagnosed systemic disease
* ≥ 5 cm (cm) (active phase) cervical dilatation
* Pregnant women who do not take any analgesia, anesthesia or anxiolytic drugs
* Spontaneous onset of labor
* Pregnant women who can speak and write Turkish well
* Pregnant woman's consent to participate in the study.

Exclusion Criteria:

* Emergency cesarean section indication
* Use of analgesic, anesthetic and anxiolytic drugs by the pregnant woman
* The pregnant woman's desire to withdraw from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — prengnancy woman
Enrollment: 45 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
paın score | pre-intervention
  Determination of pain score before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with visual pain score (0=no pain, 10=worst pain)
paın score | Between contractions within 1 hour after the intervention in the cervical dilatation range of 5-7 cm
  Determination of pain score before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with visual pain score (0=no pain, 10=worst pain)
paın score | Between contractions in about 3-4 hours after the intervention in the 8-10 cm cervical dilatation range
  Determination of pain score before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with visual pain score (0=no pain, 10=worst pain)
anxiety level | pre-intervention
  Determination of anxiety level before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with STAI From TX-I and TX-II (State-Trait Anxiety Tests) (The highest possible score is 80 and the lowest possible score is 20)
anxiety level | Between contractions within 1 hour after the intervention in the cervical dilatation range of 5-7 cm
  Determination of anxiety level before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with STAI From TX-I and TX-II (State-Trait Anxiety Tests) (The highest possible score is 80 and the lowest possible score is 20)
anxiety level | postpartum 4-24 hours
  Determination of anxiety level before and after essential oil (lemon oil and ylang ylang oil) and saline inhalation with STAI From TX-I and TX-II (State-Trait Anxiety Tests) (The highest possible score is 80 and the lowest possible score is 20)

SECONDARY OUTCOMES:
apgar score | postnatal 5. minute
  Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration." In the test, five things are used to check a baby's health. (0-10 point)
apgar score | postnatal 10. minute
  Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration." In the test, five things are used to check a baby's health. (0-10 point)

CONTACTS AND LOCATIONS:
Overall Officials: ÖZLEM ÇAĞAN, ASSİST.PROF., Study Director — Eskişehir Osmangazi University; SEVGİ KOÇ, PROF. DR., Study Director — ETLİK ZÜBEYDE HANIM GYN DISEASES TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Etlik Zübeyde Hanim Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaviani M, Maghbool S, Azima S, Tabaei MH. Comparison of the effect of aromatherapy with Jasminum officinale and Salvia officinale on pain severity and labor outcome in nulliparous women. Iran J Nurs Midwifery Res. 2014 Nov;19(6):666-72. PMID 25558267